CLINICAL TRIAL: NCT02629549
Title: A Phase 1, Single Dose, Open-Label Study to Investigate the Safety and Efficacy of OTL38 Injection for Intraoperative Imaging of Folate Receptor-alpha Positive Pituitary Adenoma
Brief Title: Intraoperative Imaging of Pituitary Adenomas by OTL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment Fulfilled
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sunil Singhal, Director, Thoracic Surgery Research Laboratory, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 822782; NCT02769533 (obsolete NCT alias)
Record Dates: First submitted 2015-12-04; First posted 2015-12-14 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Neoplasms; Pituitary Neoplasms
MeSH Terms: conditions — Neoplasms; Pituitary Neoplasms | interventions — Pafolacianine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OTL38 (Experimental): Dosage calculated by weight of individual
  Interventions: Drug: OTL38

INTERVENTIONS:
Drug: OTL38 — Infusion of OTL38 prior to surgery

SUMMARY:
The primary end-point of the study is to determine the specificity and sensitivity of OTL38 in identifying pituitary adenomas when excited by an imaging probe. The investigators intend to enroll 50 patients in this study. The study is focusing on patients presenting with suspected pituitary adenomas who are considered to be good surgical candidates.

DETAILED DESCRIPTION:
Pituitary adenomas have an estimated prevalence in the population of approximately 10%, and although they are predominantly benign tumors, they can cause significant disability from mass effect (visual field deficits and cranial nerve deficits) and from hypersecretory syndromes (Cushing's disease, acromegaly, hyperprolactinemia). Approximately 30% of all pituitary adenomas are nonfunctioning or endocrinologically silent, and despite the lack of hormonal overexpression they represent the great majority of patients of who undergo surgery given the threat of apoplexy and compression of adjacent neural structures. Surgical resection via transsphenoidal surgery remains the primary treatment modality for almost all pituitary adenomas except prolactinomas. Residual tumor, however, is quite common after surgical resection and is seen in up to 20% of surgical cases. By ensuring a negative margin through imaging during surgery, it would be possible to minimize the need for postoperative radiation therapy and/or radiosurgery and subsequent surgery as well.

Gross total resection (GTR) of a pituitary adenoma is theoretically simple but practically difficult given the intimate association of the pituitary gland with critical neurovascular structures including the internal carotid artery, optic nerves, cavernous sinus contents and adjacent frontal lobe and third ventricle. In a recent meta-analysis, functioning pituitary adenoma (Cushing's disease, prolactinoma, acromegaly) was demonstrated to have a gross total resection rate of only 78% (n=664). In another review, tabulated through multiple studies, demonstrated that for nonfunctioning pituitary adenoma, gross total resection rate ranged from 66 to 93% (n=778). Moreover, a comparison of endoscopic and microscopic removal of pituitary adenoma found the gross total resection rate was 66% using endoscopic pituitary techniques. In this context of limited ability to achieve GTR, intraoperative MRI was introduced for assessment of the degree of resection for pituitary adenoma. The intraoperative MRI is expensive, cumbersome, and impractical. A simpler means of determining the degree of resection is greatly needed in the field of brain surgery, and specifically pituitary surgery.

Pituitary adenomas are the ideal disease to investigate intra-operative imaging. Multiple studies have demonstrated that nonfunctioning pituitary adenomas express folate receptor alpha (FRα), therefore making folate receptors (FR) the ideal targets for imaging agents. While folate will initially distribute to all cells, redistribution, metabolism, and excretion will eliminate most of this agent from healthy tissues within 2-3 hours. Tumor cells that over express FRα will retain folate and any fluorescent labeled folate conjugate (such as OTL38) and internalize this.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Patients presenting with a pituitary nodule presumed to be resectable on pre-operative assessment
3. Good operative candidate
4. Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

1. Pregnant women as determined by urinary or serum beta human chorionic gonadotropin (hCG) within 72 hours of surgery
2. Patients with a history of anaphylactic reactions to OTL38
3. Patients with a known allergy to Benadryl
4. Previous exposure to OTL38

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10; Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Detection of OTL38 in tumor tissue. | 60 months
  The detection of OTL38 uptake by tumor tissue will be made with the use of an imaging system that detects the presence of dye in tissue.
Evaluate the ability of OTL38 to discern between tumorous tissue and normal, neural tissue. | 60 months
  Specificity and sensitivity of OTL38 will be calculated through the comparison of the video images gathered from the imaging system and the final pathology results from the surgical procedure.

SECONDARY OUTCOMES:
Incidence rates of all adverse events, treatment-emergent adverse events and adverse device events from time of OTL38 administration through participants' first, post-operative appointment with surgeon. | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Liu X, Ma S, Yao Y, Li G, Feng M, Deng K, Dai C, Cai F, Li Y, Zhang B, Wang R. Differential expression of folate receptor alpha in pituitary adenomas and its relationship to tumor behavior. Neurosurgery. 2012 May;70(5):1274-80; discussion 1280. doi: 10.1227/NEU.0b013e3182417e76. PMID 22089756
- [Background] Evans CO, Yao C, Laborde D, Oyesiku NM. Folate receptor expression in pituitary adenomas cellular and molecular analysis. Vitam Horm. 2008;79:235-66. doi: 10.1016/S0083-6729(08)00408-1. PMID 18804697
- [Background] Evans CO, Reddy P, Brat DJ, O'Neill EB, Craige B, Stevens VL, Oyesiku NM. Differential expression of folate receptor in pituitary adenomas. Cancer Res. 2003 Jul 15;63(14):4218-24. PMID 12874029
- [Background] Feng Y, Shen J, Streaker ED, Lockwood M, Zhu Z, Low PS, Dimitrov DS. A folate receptor beta-specific human monoclonal antibody recognizes activated macrophage of rheumatoid patients and mediates antibody-dependent cell-mediated cytotoxicity. Arthritis Res Ther. 2011 Apr 8;13(2):R59. doi: 10.1186/ar3312. PMID 21477314
- [Background] Hilgenbrink AR, Low PS. Folate receptor-mediated drug targeting: from therapeutics to diagnostics. J Pharm Sci. 2005 Oct;94(10):2135-46. doi: 10.1002/jps.20457. PMID 16136558
- [Background] Kennedy MD, Jallad KN, Thompson DH, Ben-Amotz D, Low PS. Optical imaging of metastatic tumors using a folate-targeted fluorescent probe. J Biomed Opt. 2003 Oct;8(4):636-41. doi: 10.1117/1.1609453. PMID 14563201
- [Background] Low PS, Antony AC. Folate receptor-targeted drugs for cancer and inflammatory diseases. Adv Drug Deliv Rev. 2004 Apr 29;56(8):1055-8. doi: 10.1016/j.addr.2004.02.003. No abstract available. PMID 15094205
- [Background] Xia W, Low PS. Folate-targeted therapies for cancer. J Med Chem. 2010 Oct 14;53(19):6811-24. doi: 10.1021/jm100509v. No abstract available. PMID 20666486
- [Background] Lu Y, Sega E, Leamon CP, Low PS. Folate receptor-targeted immunotherapy of cancer: mechanism and therapeutic potential. Adv Drug Deliv Rev. 2004 Apr 29;56(8):1161-76. doi: 10.1016/j.addr.2004.01.009. PMID 15094213
- [Background] Lu Y, Xu LC, Parker N, Westrick E, Reddy JA, Vetzel M, Low PS, Leamon CP. Preclinical pharmacokinetics, tissue distribution, and antitumor activity of a folate-hapten conjugate-targeted immunotherapy in hapten-immunized mice. Mol Cancer Ther. 2006 Dec;5(12):3258-67. doi: 10.1158/1535-7163.MCT-06-0439. PMID 17172429
- [Background] Paulos CM, Reddy JA, Leamon CP, Turk MJ, Low PS. Ligand binding and kinetics of folate receptor recycling in vivo: impact on receptor-mediated drug delivery. Mol Pharmacol. 2004 Dec;66(6):1406-14. doi: 10.1124/mol.104.003723. Epub 2004 Sep 15. PMID 15371560
- [Background] Stephenson SM, Low PS, Lee RJ. Folate receptor-mediated targeting of liposomal drugs to cancer cells. Methods Enzymol. 2004;387:33-50. doi: 10.1016/S0076-6879(04)87003-4. No abstract available. PMID 15172156
- [Background] Yang J, Chen H, Vlahov IR, Cheng JX, Low PS. Characterization of the pH of folate receptor-containing endosomes and the rate of hydrolysis of internalized acid-labile folate-drug conjugates. J Pharmacol Exp Ther. 2007 May;321(2):462-8. doi: 10.1124/jpet.106.117648. Epub 2007 Feb 8. PMID 17289839
- [Background] Dorward NL. Endocrine outcomes in endoscopic pituitary surgery: a literature review. Acta Neurochir (Wien). 2010 Aug;152(8):1275-9. doi: 10.1007/s00701-010-0649-y. Epub 2010 May 10. PMID 20454982
- [Background] Swearingen B. Update on pituitary surgery. J Clin Endocrinol Metab. 2012 Apr;97(4):1073-81. doi: 10.1210/jc.2011-3237. Epub 2012 Feb 15. PMID 22337908
- [Background] Berkmann S, Schlaffer S, Nimsky C, Fahlbusch R, Buchfelder M. Follow-up and long-term outcome of nonfunctioning pituitary adenoma operated by transsphenoidal surgery with intraoperative high-field magnetic resonance imaging. Acta Neurochir (Wien). 2014 Dec;156(12):2233-43; discussion 2243. doi: 10.1007/s00701-014-2210-x. Epub 2014 Sep 2. PMID 25174805
- [Background] Sylvester PT, Evans JA, Zipfel GJ, Chole RA, Uppaluri R, Haughey BH, Getz AE, Silverstein J, Rich KM, Kim AH, Dacey RG, Chicoine MR. Combined high-field intraoperative magnetic resonance imaging and endoscopy increase extent of resection and progression-free survival for pituitary adenomas. Pituitary. 2015 Feb;18(1):72-85. doi: 10.1007/s11102-014-0560-2. PMID 24599833